CLINICAL TRIAL: NCT04458818
Title: A Novel Approach for Thyroplasty Type 1, With Prolene Mesh. A Prospective Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Rashid (Other)
Responsible Party: Sponsor-Investigator, Muhammad Rashid, Professor of ENT, Pak Emirates Military Hospital
Organization: Pak Emirates Military Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prolene mesh VC medialization
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Vocal Cord Paralysis; Phonasthenia; Presbylarynges; Idiopathic Vocal Cord Paralysis; Ca Larynx
Keywords: Voice Rehabilitation; Vocal Medialization; Prolene mesh implant
MeSH Terms: conditions — Vocal Cord Paralysis; Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: The single group will be implanted with Prolene mesh made into Swiss rolls and placed in Laryngeal Window between the cartilage and inner periosteum,
Masking Description: No Masking. Patients in one arm are provided with prolene mesh implant, and is known by the patient, health care provider and the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolene Mesh Implant (Experimental): The Group of Patients who were offered Prolene mesh Laryngeal implants for Vocal Cord Medialization.
  Interventions: Procedure: Prolene Mesh Vocal Cord Medialization Implant

INTERVENTIONS:
Procedure: Prolene Mesh Vocal Cord Medialization Implant — The surgery will be performed under local anesthesia (lignocaine with adrenaline 2%) and procedural sedation with propofol 25-100mcg/kg/min (only sedative dose) will be administered, so that the patient remains vocally responsive during the procedure. Incision will be made at the lower border of thyroid cartilage under aseptic measures. Skin flaps will be raised in sub-platysmal plane, strap muscles will be separated in the midline to expose the laryngeal cartilaginous framework. A simple laryngeal window approach will be used to place the Ethicon prolene mesh 6 x 6cm Swiss roll, secured with prolene 2/0 suture trimmed to the required size. Post op voice analysis will be done on 7th day and 14th post-operative day. Monthly follow up will be advised after that.

SUMMARY:
Larynx performs important functions of the aero-digestive tract, it has vital role in control of breathing, phonation, deglutition and protection of lower respiratory tract from aspiration. Vocal cord paralysis is a common and at times debilitating laryngeal dysfunction that has great social and economic impact on patients life. Medialization thyroplasty (MT), if done accurately and up to the expectations of the patient is very rewarding. However different materials with some modifications in the technique of the classical Isshiki type 1 thyroplasty is in practice, each with its own profile of benefits and disadvantages. Most of them are costly and out of reach of general population. In this regard, we aim to test a prolene mesh implant, which is easily available and can be placed with relative ease.

DETAILED DESCRIPTION:
Introduction: Larynx performs important functions of the aero-digestive tract, it has vital role in control of breathing, phonation, deglutition and protection of lower respiratory tract from aspiration. The function of Vocal cord is central to all the Laryngeal functions, even unilateral paralysis can have profound effect on overall laryngeal functionality especially in sound production. Around 80% of all the jobs in the world are somehow dependent upon social communication. Vocal cord paralysis is a common and at times debilitating laryngeal dysfunction that has great social and economic impact on patients life. Medialization thyroplasty (MT), if done accurately and up to the expectations of the patient is very rewarding. However different materials with some modifications in the technique of the classical Isshiki type 1 thyroplasty is in vogue, each with its own profile of benefits and disadvantages. In this regard a large variety of complex materials are in use, which are not routinely available in developing countries and some of them have not been cleared by the host countries medical authorities. Most of them are costly and out of reach of general population. In this regard, we aim to test a prolene mesh implant, which is easily available and can be placed with relative ease. We recommend some modifications in the original technique, which would not require the complex measurements and costly equipment. Even it can be performed without fiber-optic laryngoscope guidance. Prolene is already in use in wide range of procedures worldwide, approved by Federal drug administration in 1997 but it has never been used in larynx. We intend to explore the efficacy of prolene mesh as an implant for vocal cord medialization in terms of patient satisfaction and voice outcome.

Objective: To evaluate a new approach of vocal cord medialization using prolene mesh as an implant material.

Study Design: Interventional, prospective study.. Place and Duration of study: Ent departments of multiple tertiary care hospitals of Pakistan from Jun 2020 and onwards.

Materials and Methods: Patients of age 15 years onwards and with vocal cord paralysis/ paresis due to multiple causes would included in the study. Patients with neoplasm, trauma and underlying muscular dystrophy are to be excluded. All patients will be counselled properly and given the choice of intervention by prolene mesh implant. Consenting patients will be subjected to routine blood investigations with fiber optic laryngoscopy and imaging with Computerized Tomography scan (where applicable). Procedure will be performed under local anesthesia with mild sedation, so that the patient will remain vocally responsive for the assessment of voice and breathing intraoperatively. Pre and postoperative voices will be recorded with a standard microphone at 15cm distance from the mouth in a quiet room. Maximum phonation time (MPT) while vocalizing the vowel sound 'eee' and Maximum words count (MWC) in a single breath (counting numbers) will be recorded pre and post operatively. Maximum three attempts will be allowed to each patient and the better score of the three will be recorded in the data. For subjective assessment of voice quality Visual (1-10) analogue score (VAS) will be used both pre and postoperatively. For objective assessment of patients a customized Voice Handicap Index (VHI-10) will be used.

Modified VHI-10 Questionnaire

1. My voice makes it difficult for people to hear me. 0 1 2 3 4 5
2. I run out of air when I talk. 0 1 2 3 4 5
3. People have difficulty understanding me in noisy room. 0 1 2 3 4 5
4. I use a great deal of effort to speak. 0 1 2 3 4 5
5. My family has difficulty hearing me when I call them throughout the house. 0 1 2 3 4 5
6. I use phone less often than I would like to. 0 1 2 3 4 5
7. I am tense when I am talking to others because of my voice. 0 1 2 3 4 5
8. I tend to avoid groups of people because of my voice. 0 1 2 3 4 5
9. People seem irritated with my voice. 0 1 2 3 4 5
10. People ask what's wrong with my voice. 0 1 2 3 4 5 VHI : Voice Handicap Index 0 = never, 1 = almost never (occasionally), 2 = sometimes, 3 = almost always, 4 = always Fig 1.1 Modified Voice Handicap Index (VHI-10)

Hospital ethical committee's approval will be obtained. The surgery will be performed under local anesthesia (lignocaine with adrenaline 2%) and procedural sedation with propofol 25-100mcg/kg/min (only sedative dose) will be administered, so that the patient remains vocally responsive during the procedure. Incision will be made at the lower border of thyroid cartilage under aseptic measures. Skin flaps will be raised in sub-platysmal plane, strap muscles will be separated in the midline to expose the laryngeal cartilaginous framework. A simple laryngeal window approach will be used to place the Ethicon prolene mesh 6 x 6 cm Swiss roll, secured with prolene 2/0 suture trimmed to the required size. Post op voice analysis will be done on 14th post-operative day. Routine monthly follow up for 3 months will be advised after that.

The results will be analyzed using Internal IBM SPSS Statistics version 20. Variables defined would be compared between the preoperative and postoperative groups. For normal data paired sample t-test would be used and for abnormally distributed data non parametric t-test would be used. P-value of less than 0.05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 15 years
* Vocal cord paralysis

Exclusion Criteria:

* Patients with neoplasms
* Trauma
* Muscular dystrophies

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ENT Departments, Kharian, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 01 May 2020 - 30 Jan 2021
Pre-assignment Details: Before inducting into the study, patients were tested with exclusion criteria i.e Neoplasia, trauma and muscular dystrophy cases, and inclusion criteria i.e.15 years and younger, vocal cord paralysis and voice disability.
Period: Overall Study
Arm/Group | Prolene Mesh Implant
Started | 39 (May 01 2020)
Completed | 39 (Jan 30 2021)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prolene Mesh Implant
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 32
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Phonation Time
Description: Pre and postoperative voices will be recorded with a standard microphone at 15cm distance from the mouth in a quiet room. Maximum phonation time (MPT) while vocalizing the vowel sound 'eee' will be measured in seconds. Maximum three attempts will be allowed to each patient and the better score of the three will be recorded in the data.
Time Frame: Preoperative and 14th Postoperative day
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Prolene Mesh Implant
Number analyzed (Participants) | 39
seconds
  pre operative | 7.74 (1.712)
  post operative | 14.08 (3.390)

2. Primary Outcome: Change in Maximum Words Count
Description: Pre and postoperative voices will be recorded with a standard microphone at 15cm distance from the mouth in a quiet room. Maximum words count (MWC) in a single breath (counting numbers) will be recorded pre and post operatively. Maximum three attempts will be allowed to each patient and the better score of the three will be recorded in the data.
Time Frame: Preoperative and 14th Postoperative day
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Prolene Mesh Implant
Number analyzed (Participants) | 39
words
  pre operative | 11.33 (3.359)
  post operative | 18.28 (5.047)

3. Primary Outcome: Change in Voice Quality on Visual Analogue Score
Description: For subjective assessment of voice quality Visual (1-10) analogue score (VAS) will be used both pre and postoperatively. Score 1 will be the score for lowest and 10 being the best score for voice quality.
Time Frame: Preoperative and 14th Postoperative day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prolene Mesh Implant
Number analyzed (Participants) | 39
score on a scale
  pre operative | 4.77 (1.224)
  post operative | 7.64 (1.308)

ADVERSE EVENTS:
Time Frame: 1 year follow up was kept for all the patients.
Arm/Group | Prolene Mesh Implant
All-Cause Mortality (participants affected / at risk) | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 5/39
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prolene Mesh Implant (N=39)
URTI (Respiratory, thoracic and mediastinal disorders) | 4 (39) — Upper respiratory tract infections
skin infection (Infections and infestations) | 1 (39) — Wound infection, post operatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT04458818/Prot_SAP_000.pdf